CLINICAL TRIAL: NCT02915068
Title: Feasibility of a Clinician Training Program to Improve Patient-provider Communication in the Presence of Health IT Systems in the Exam Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Minal Patel, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HUM00100232
Record Dates: First submitted 2016-09-20; First posted 2016-09-26 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: patient-provider communication; Electronic Health Records; Provider education
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Physicians do not receive focused education and training on patient-centered communication with the EHR
- EHR-PACE (Experimental): participants will receive EHR-PACE, an interactive 1.5 hour training module that teaches clinicians best practices for communicating with patients in the presence of computer systems in the exam room (specifically EHRs).
  Interventions: Behavioral: EHR-Physician Asthma Care Education Program

INTERVENTIONS:
Behavioral: EHR-Physician Asthma Care Education Program — participants will receive EHR-PACE, an interactive 1.5 hour training module that teaches clinicians best practices for communicating with patients in the presence of computer systems in the exam room (specifically EHRs).
  Arms: EHR-PACE

SUMMARY:
The investigators propose to modify and expand the internationally-recognized evidence-based Physician Asthma Care Education (PACE) program to make it a suitable tool for training primary care clinicians on the effective use of EHRs at the point of care. The investigators will first develop the EHR edition of PACE (EHR-PACE) through literature and expert review of best practices for clinicians interacting with patients in the presence of computer systems in the exam room. They will then establish the feasibility and potential impact of EHR-PACE via a randomized design on 125 patients of 20 physicians who receive the intervention on the following outcomes via survey 3 and 6 months post-intervention: patient satisfaction with the physician's performance, asthma control, and asthma-related quality of life. Outcomes will be assessed on patients, but physicians will receive the intervention. Patients will not know which arm their doctor was randomized to. The pilot trial will compare two groups of primary care physicians who see patients with asthma in clinics equipped with certified EHRs. It is hypothesized that patients of physicians who receive EHR-PACE training will achieve better outcomes compared to physicians who do not receive EHR-PACE.

DETAILED DESCRIPTION:
Failure in clinician-patient communication, lack of clarity regarding clinical treatment priorities, and more recently, ineffective use of health IT systems in exam rooms are associated with deficits in achieving chronic disease management goals, and increased healthcare utilization and costs. Strategies for communicating with patients in exam rooms in the presence of electronic health records (EHR) have been described in the literature. Whether such strategies are reaching clinicians and demonstrating positive health outcomes is unclear. The investigators propose to develop and test the feasibility on patient outcomes of an interactive training module that teaches clinicians best practices for communicating with patients in the presence of computer systems in the exam room (specifically EHRs). They propose to modify and expand the internationally-recognized evidence-based Physician Asthma Care Education (PACE) program to make it a suitable tool for training primary care clinicians on the effective use of EHRs at the point of care. The PACE program is based on concepts and skills for strengthening communication and patient-clinician relationships through behavior change principles that are highly applicable to patients with asthma and has potential for specific application to EHR use in clinical practice. The investigators will first develop the EHR edition of PACE (EHR-PACE) through literature and expert review of best practices for clinicians interacting with patients in the presence of computer systems in the exam room. They will then establish the feasibility and potential impact of EHR-PACE via a randomized design on 125 patients of 20 physicians who receive the intervention on the following outcomes via survey 3 and 6 months post-intervention: patient satisfaction with the physician's performance, asthma control, and asthma-related quality of life. Outcomes will be assessed on patients, but physicians will receive the intervention.Patients will not know which arm their doctor was randomized to.The pilot trial will compare two groups of primary care physicians who see patients with asthma in clinics equipped with certified EHRs. It is hypothesized that patients of physicians who receive EHR-PACE training will achieve better outcomes compared to physicians who do not receive EHR-PACE.

EHR-PACE developed in this study is expected to have a high degree of relevance for improving the patient-provider communication skills of clinicians who see a wide range of patients in a variety of practice settings that have now integrated EHRs. Given that PACE can achieve dramatic outcomes within only two, 2-hour sessions, EHR-PACE has the potential to become an invaluable training tool to busy clinicians if proven feasible and effective. Ultimately, this work has potential for a high degree of impact.

ELIGIBILITY:
Inclusion Criteria:

Physicians:

1. Licensed physician in practice and board certified in primary care or family medicine
2. Treating adults with asthma
3. Full-time in a practice at an Integrated Health Associates clinic that has implemented a certified EHR system for at least one year
4. Consent to participate
5. Will generate a roster of adult asthma patients for inclusion in the study

Patients:

1. Treated by the participating physician during the study intake period
2. 18 years of age or older
3. Have a diagnosis of asthma made by a physician using the National Asthma Education and Prevention Program Guidelines
4. Have at least one urgent medical care visit for asthma in the previous year
5. Have access to a telephone
6. Consent to participate

Exclusion Criteria:

Patients:

1. Have other chronic disorders that have pulmonary complications

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-06; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline patient report of physician performance at 3 and 6 months | baseline, 3 months, 6 months
  The patient's report of physician performance will be used as the key measure in this study. They will use a validated instrument previously developed by the research group in the PACE trials, focusing on clinical practices of the clinician, especially, use of National Asthma Education and Prevention Program recommended therapies, communication and counseling behaviors specially related to EHR use.

SECONDARY OUTCOMES:
Change from baseline patient satisfaction at 3 and 6 months | baseline, 3 months, 6 months
  specific facets of satisfaction with care adapted from the widely used Patient Satisfaction Questionnaire, especially as it relates to interactions with clinicians in the presence of EHRs in the exam room
Change from baseline asthma control at 3 and 6 months | baseline, 3 months, 6 months
  the Asthma Control Test (ACT), a valid measure responsive to changes in asthma control over time
Change from baseline asthma-related quality of life at 3 and 6 months | baseline, 3 months, 6 months
  Mini Asthma Quality of Life Questionnaire (Mini-AQLQ), a 15-item validated instrument that assesses physical, emotional, and social well-being of adults with asthma through four domains (activity limitations, symptoms, emotional function, and exposure to environmental stimuli).

CONTACTS AND LOCATIONS:
Overall Officials: Minal R Patel, PhD, MPH, Principal Investigator — Assistant Professor
Locations (1):
- Integrated Health Associates ClinSite Research, Ann Arbor, Michigan, United States